CLINICAL TRIAL: NCT06265233
Title: Pilot Study of Cognitive Behavioral Therapy (CBT) Plus Improv Group Therapy for OCD
Brief Title: ERP Plus Improv Group Therapy for OCD (IMPROVE Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69668
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Behavioral Therapy; ExRP (Exposure and Response Prevention); ERP; Improv comedy; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERP combined with Improv Group Therapy (Experimental): Participants will attend 90-minute ERP + improv group therapy sessions for 12 consecutive weeks. They will also complete homework between sessions, answer questions, and complete questionnaires.
  Interventions: Other: Group Improv sessions; Behavioral: Group Exposure and Response Prevention (ERP) Therapy

INTERVENTIONS:
Other: Group Improv sessions — Therapist-led 90-minute exposure and response prevention (ERP) combined with improv sessions.
  Other Names: Improv Comedy
Behavioral: Group Exposure and Response Prevention (ERP) Therapy — Therapist-led 90-minute exposure and response prevention (ERP) combined with improv sessions.
  Other Names: ERP

SUMMARY:
The goal of this study is to pilot test a novel group therapy intervention for adults with OCD.

DETAILED DESCRIPTION:
The intervention will incorporate exposure and response prevention (ERP) with improvisational comedy ("improv") activities. ERP is the gold-standard treatment for OCD. Improv comedy is a type of theater in which actors perform without a script. This study aims to evaluate whether the intervention is helpful for reducing OCD symptoms and intolerance of uncertainty (a mechanism maintaining OCD). It will also explore whether the intervention is feasible and acceptable.

During the group therapy sessions, participants will engage with improv comedy exercises that have been adapted to function as exposures for different types of OCD. Participants will:

* attend an ERP + improv group therapy intervention (90-minute sessions for 12 weeks)
* complete homework in-between sessions
* answer questions
* complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to speak and understand English
* Clinical diagnosis of obsessive-compulsive disorder (OCD)

Exclusion Criteria:

* Current active suicidality
* Medical or psychiatric illness that could interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Change in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline and up to 12 weeks
  Change in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% change on the YBOCS.

SECONDARY OUTCOMES:
Change in Intolerance of Uncertainty Score | Baseline and up to 12 weeks
  Change in intolerance of uncertainty (IU) will be measured with the Intolerance of Uncertainty Scale - Short Form (IUS-12). IU is the tendency to respond negatively to uncertain situations. The IUS-12 is a 12-item self-report measure that assesses IU. Each item is assessed using a 5-point Likert scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me).
  It consists of two subscales: Prospective IU and Inhibitory IU. Prospective IU is the cognitive appraisal of a threat related to future uncertainty. Inhibitory IU refers to the behavioral inhibition related to uncertainty. The Prospective IU subscale is comprised of 7 items, while the Inhibitory IU subscale is comprised of 5 items. Scores are summed to generate the two subscale scores and a total score. Total IUS-12 scores range from 12 to 60, with higher scores indicating a higher IU.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- 401 Quarry, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford OCD Research Lab Website — https://med.stanford.edu/rodriguezlab/research.html